CLINICAL TRIAL: NCT07233902
Title: Comparison of the Effects of Synchronous and Asynchronous Exercise Programs in Patients With Multiple Sclerosis
Brief Title: MS Synchronous vs Asynchronous Exercise Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yeditepe University (Other)
Collaborators: The Scientific and Technological Research Council of Turkey (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: YEDITEPE-MS-SYNCASYNC-2025; TUBITAK 1002-A 125S054 (Other Grant/Funding Number: TUBITAK)
Record Dates: First submitted 2025-11-13; First posted 2025-11-18 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2025-11

CONDITIONS: Multiple Sclerosis; Multiple Sclerosis (MS) - Relapsing-remitting
Keywords: multiple sclerosis; online exercise; tele-rehabilitation; synchronous; asynchronous
MeSH Terms: conditions — Multiple Sclerosis; Multiple Sclerosis, Relapsing-Remitting

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Outcome assessors were blinded to group allocation. Participants and intervention providers were aware of group assignments due to the nature of the intervention delivery (synchronous vs asynchronous).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Synchronous Exercise Group (Experimental): Participants in this group receives a 12-week structured exercise program delivered synchronously twice per week through live online video sessions (Google Meet or WhatsApp). Each session lasts approximately 40 minutes and included 10 minutes of warm-up, 25 minutes of strengthening and core stabilization exercises, and 5 minutes of cool-down stretching. All sessions are supervised in real time by a physiotherapist.
  The program focuses on improving functional capacity, muscle strength, fatigue, independence, and quality of life in individuals with relapsing-remitting multiple sclerosis.
  Interventions: Other: Combined Exercise Program (Synchronous Delivery)
- Asynchronous Exercise Group (Active Comparator): Participants in this group receives the same 12-week structured exercise program delivered asynchronously through pre-recorded videos shared online twice per week. Each session lasts approximately 40 minutes, including warm-up, main strengthening/core exercises, and cool-down.
  Participants maintain exercise logs and reported adherence weekly. Physiotherapists monitor logs and provided feedback via e-mail or phone as needed. The program targets the same outcomes as the synchronous intervention.
  Interventions: Other: Combined Exercise Program (Asynchronous Delivery)

INTERVENTIONS:
Other: Combined Exercise Program (Synchronous Delivery) — Participants receive a 12-week structured combined exercise program delivered twice weekly via live online video sessions (Google Meet or WhatsApp). Each session lasts approximately 40 minutes and included 10 minutes of warm-up, 25 minutes of strengthening and core stabilization exercises, and 5 minutes of cool-down stretching.
  Exercise intensity is maintained between 12 and 15 on the Borg Rating of Perceived Exertion scale. Rest periods are adjusted individually. Exercises are supervised in real time by a physiotherapist, who monitored participants' form, safety, and perceived fatigue throughout each session
  Arms: Synchronous Exercise Group
Other: Combined Exercise Program (Asynchronous Delivery) — Participants follow the same 12-week structured exercise program twice weekly using pre-recorded instructional videos. The program consists of warm-up, strengthening/core, and cool-down components identical to the synchronous arm.
  Participants receive detailed guidance to ensure correct posture and performance, logged each session in exercise diaries, and submitted weekly feedback to researchers. Investigators review exercise logs and provided individualized feedback via e-mail or phone. In case of difficulties, participants can contact the research team for assistance
  Arms: Asynchronous Exercise Group

SUMMARY:
This randomized controlled study aims to compare the effects of synchronous and asynchronous exercise programs on individuals diagnosed with relapsing-remitting multiple sclerosis (RRMS). Participants meeting the inclusion criteria (EDSS score between 2 and 5.5, aged 18-55) were randomly assigned to either the Synchronous Exercise Group (SEG) or the Asynchronous Exercise Group (ASEG).

The synchronous program was delivered via live online sessions using Google Meet and WhatsApp video calls, while the asynchronous program consisted of pre-recorded exercise videos accessible to participants. Both programs included structured exercises focusing on functional capacity, muscle strength, fatigue, independence, and quality of life.

The sample size was determined using G*Power software based on previous studies in individuals with multiple sclerosis, targeting a total of 16. Statistical analyses will be conducted using SPSS 26.0. Parametric and non-parametric tests will be used depending on data distribution, with significance set at p < 0.05.

The study seeks to improve accessibility to exercise programs for MS patients and provide evidence for the efficacy of remotely delivered synchronous versus asynchronous rehabilitation models.

DETAILED DESCRIPTION:
This randomized controlled trial was designed to evaluate and compare the effects of synchronous and asynchronous structured exercise programs in individuals diagnosed with relapsing-remitting multiple sclerosis (RRMS). The main aim was to investigate differences in fatigue, functional exercise capacity, muscle strength, functional independence, and quality of life between the two intervention models.

Participants were recruited according to the inclusion criteria: age 18-55, RRMS diagnosis according to McDonald criteria, Expanded Disability Status Scale (EDSS) score between 2 and 5.5, no relapse within the last six months, and access to technological infrastructure (internet, camera, microphone). Exclusion criteria included other neurological diagnoses, cardiovascular, vestibular, or orthopedic conditions limiting exercise participation, cognitive impairment (Mini-Mental State Examination <24), fall risk (Timed Up and Go >14.2 s), psychiatric disorders, vision or hearing impairments, pregnancy, or concurrent physiotherapy programs.

Participants were randomly assigned into two groups (n=20 each): the Synchronous Exercise Group (SEG) and the Asynchronous Exercise Group (ASEG). Both groups performed a 12-week combined exercise program (2 sessions per week, 40 minutes per session) consisting of strengthening, core stabilization, and respiratory exercises, followed by a 3-month follow-up period. The structured program included warm-up (10 min: rhythmic stepping, diaphragmatic breathing, shoulder mobility), main exercises (25 min: bridging, plank, squats, seated upper-limb strengthening), and cool-down (5 min: stretching and relaxation).

The synchronous group performed exercises live through Google Meet or WhatsApp video calls under real-time physiotherapist supervision. The asynchronous group followed pre-recorded video sessions and submitted exercise logs weekly; feedback and follow-up were provided via e-mail or phone.

Assessments were conducted at four time points: baseline (D0), mid-intervention (4th week; D1), post-intervention (12th week; D2), and after a 3-month follow-up (D3). Statistical analyses were performed using SPSS 26.0; normality was assessed via the Kolmogorov-Smirnov test. Within-group comparisons used paired-sample t tests or Wilcoxon tests, and between-group differences were analyzed using independent t tests or Mann-Whitney U tests. Repeated-measures ANOVA was applied for follow-up analyses, with significance set at p < 0.05.

The study hypothesized that synchronous telerehabilitation would result in superior outcomes compared to asynchronous exercise delivery in terms of fatigue reduction, muscle strength improvement, and enhanced functional capacity.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Relapsing-Remitting Multiple Sclerosis (RRMS) according to the McDonald criteria.
* Age between 18 and 55 years.
* Expanded Disability Status Scale (EDSS) score between 2.0 and 5.5.
* No relapse within the last six months.
* Access to the necessary technological infrastructure (internet, camera, and microphone) to participate in the synchronous exercise program.

Exclusion Criteria:

* Presence of any neurological diagnosis other than MS.
* Any vestibular, cardiovascular, or orthopedic condition that limits exercise participation or increases fall risk (Jallouli et al., 2022).
* Mini-Mental State Examination (MMSE) score below 24.
* Timed Up and Go (TUG) test result greater than 14.2 seconds, indicating elevated fall risk (Block et al., 2022).
* Severe visual or auditory impairments.
* Presence of a psychiatric diagnosis.
* Current participation in another exercise or physiotherapy/rehabilitation program.
* Pregnancy.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2025-04-01 (Actual); Primary Completion 2025-10-01 (Actual); Study Completion 2025-10-29 (Actual)

PRIMARY OUTCOMES:
6 Minute Walk Test | 24 weeks
  The 6-Minute Walk Test is a submaximal functional exercise test used to evaluate aerobic capacity, endurance, and functional mobility in individuals with multiple sclerosis.
Respiratory Muscle Strength | 24 weeks
  Respiratory muscle strength is assessed through Maximal Inspiratory Pressure and Maximal Expiratory Pressure measurements obtained with a MicroRPM Pressure Meter. Participants are instructed to place the mouthpiece in their mouth while using a nose clip to prevent air leakage.
Fatigue Severity Scale | 24 weeks
  The Fatigue Severity Scale evaluates the impact and severity of fatigue in daily life activities, particularly in individuals with neurological conditions such as multiple sclerosis.
Multiple Sclerosis Quality of Life Scale | 24 weeks
  The Multiple Sclerosis Quality of Life Scale is a disease-specific health-related quality of life instrument for individuals with multiple sclerosis. The subscales include physical function, role limitations due to physical problems, pain, emotional well-being, energy, health perceptions, social function, cognitive function, health distress, sexual function, overall quality of life, and satisfaction with sexual function.
Five Times Sit-to-Stand Test | 24 weeks
  The Five Times Sit-to-Stand Test is a simple and reliable clinical measure used to assess lower limb muscle strength, functional mobility, and fall risk in individuals with multiple sclerosis.

SECONDARY OUTCOMES:
Beck Depression Inventory | 24 weeks
  The Beck Depression Inventory is a self-report scale designed to measure the severity of depressive symptoms. The inventory consists of 21 items, each rated on a 4-point Likert scale.
Beck Anxiety Inventory | 24 weeks
  The Beck Anxiety Inventory measures the frequency and severity of anxiety symptoms experienced during the past week. The instrument contains 21 items, each rated on a 4-point scale (0-3), from "not at all" to "severely." The total score ranges from 0 to 63, where higher scores indicate higher anxiety.
Montreal Cognitive Assessment | 24 weeks
  The Montreal Cognitive Assessment was developed by Nasreddine et al. (2005) to detect mild cognitive impairment. It evaluates multiple cognitive domains including visuospatial/executive skills, naming, memory, attention, language, abstraction, delayed recall, and orientation.
Berg Balance Scale | 24 weeks
  The Berg Balance Scale is a performance-based measure of static and dynamic balance. The scale includes 14 items, each scored from 0 (unable to perform) to 4 (performs independently), yielding a maximum total score of 56.
Dynamic Gait Index | 24 weeks
  The Dynamic Gait Index assesses dynamic balance, gait adaptability, and fall risk during walking under various conditions. It consists of 8 tasks, such as level walking, changing speed, head turns, stepping over and around obstacles, pivot turns, and stair negotiation.

CONTACTS AND LOCATIONS:
Locations (1):
- Yeditepe University, Istanbul, Ataşehir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared publicly due to ethical and privacy considerations. Group-level results, aggregated data, and summary analyses may be shared upon reasonable request from qualified researchers after publication of the main study findings.